CLINICAL TRIAL: NCT02701231
Title: Low-frequency Rotating Magnetic System Combined With Systemic Anti-tumor Therapy for Advanced Lung Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese PLA General Hospital (Other)
Collaborators: Xijing Hospital (Other); Shandong University of Traditional Chinese Medicine (Other); Shandong Provincial Hospital (Other Government)
Responsible Party: Principal Investigator, Chen Liang_An, Director of respiratory medicine, Chinese PLA General Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: S2015-093-01
Record Dates: First submitted 2016-01-20; First posted 2016-03-08 (Estimated); Last update posted 2016-03-09 (Estimated); Status verified 2016-03

CONDITIONS: Lung Neoplasms
Keywords: lung cancer; Low-frequency rotating magnetic therapy system; systemic anti-tumor therapy
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sham control (Sham Comparator): Subjects will receive one cycle of treatment of sham low-frequency rotating magnetic therapy system plus systemic anti-tumor therapy after randomization
  Interventions: Drug: Systemic anti-tumor therapy; Device: Sham Low-frequency Rotating Magnetic Therapy System
- Low-frequency Rotating Magnetic Therapy (Experimental): Subjects will receive one cycle of treatment of low-frequency rotating magnetic therapy system plus systemic anti-tumor therapy after randomization
  Interventions: Device: Low-frequency Rotating Magnetic Therapy System; Drug: Systemic anti-tumor therapy

INTERVENTIONS:
Device: Low-frequency Rotating Magnetic Therapy System — Two pairs of fan-shaped NdFeB permanent magnets were attached to a circular iron plate and arranged to establish magnetic field. The bottom two magnets rotated at certain frequency driven by a step motor, which was controlled using a functional signal generator. The top two magnets rotated synchronously due to the strong magnetic interaction. Magnetic flux density was measured at the target site using a gauss meter. The entire magnetic apparatus was located in a hood with humidity and temperature controller.
  Arms: Low-frequency Rotating Magnetic Therapy
Drug: Systemic anti-tumor therapy — Systemic anti-tumor therapy includes targeted therapies, chemotherapy and best supportive care, according to NCCN non-small cell lung cancer(NSCLC) and small cell lung cancer(SCLC) guidelines. SCLC patients will receive six cycles of cisplatin and etoposide. NSCLC patients will receive EGFR and ALK test. With sensitive result the first-line therapy will be Erlotinib/Gefitinib/Crizotinib. If insensitive, the patient will receive six cycles of cisplatin and pemetrexed. Then the patient will receive tumor response evaluation. The patient with response or stable disease will receive maintenance therapy with one or some of the drugs including bevacizumab, pemetrexed, gemcitabine and docetaxel until disease progression. During experience all patients will receive clinical observation. Once proven for disease progression the patient will finish the experiment.
  Other Names: Systemic therapies for advanced lung cancer
Device: Sham Low-frequency Rotating Magnetic Therapy System — Sham Low-frequency Rotating Magnetic Therapy System is a similar apparatus except that there were two rotating iron plates instead of magnets, thus lacking a magnetic field.
  Arms: Sham control

SUMMARY:
The purpose of this study is to determine whether Low-frequency Rotating Magnetic Therapy System is effective and safe in the treatment of advanced lung cancer.

DETAILED DESCRIPTION:
The purpose of this study is to assess the efficacy and safety of the Low-frequency Rotating Magnetic Therapy System(with systemic anti-tumor therapy) compared to systemic anti-tumor therapy in patients suffering from advanced lung cancer.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to give written informed consent
* Male or female aged 18 years and older
* Histologic diagnosis of non-small cell lung cancer (unable to receive surgery) or small cell lung cancer (limited stage or extensive stage)
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) ≤ 3- going to receive systemic anti-tumor therapy
* Measurable disease based on RECIST 1.1
* Adequate hematologic and organ function

Exclusion Criteria:

* Currently participating and receiving study therapy in, or has participated in a study of an investigational agent and received study therapy or used an investigational device
* Unable to lie in bed
* With any metal implants in body
* Human immunodeficiency virus (HIV)
* Malignancies other than lung cancer within 5 years prior to randomization
* History or current evidence of any condition, therapy or laboratory abnormality that might confound the results of the trial or interfere with the subject's participation for the full duration of the trial
* Pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2015-11; Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Functional Assessment of Cancer Therapy-Lung Questionaire（FACT-L） | within six weeks after randomization
  Use the FACT-L to assess the effiency of low-frequency rotating magnetic system on the improvement of patients' quality of life
Number of Participants With Adverse Events That Are Related to Treatment | From first time of study treatment until 90 days after the last, assessed up to 4 months
  AEs: Type, incidence, severity, seriousness and relationship to study medications of adverse events (AE) (graded by the National Cancer Institute [NCI] Common Terminology Criteria for Adverse Events [CTCAE 4.0]

SECONDARY OUTCOMES:
Duration of response according to standard RECIST v1.1 | up to 5 years after the first patient randomized
  At each visit subjects will be programmatically assigned a RECIST visit response of CR, PR, SD or PD depending on the status of their disease compared to baseline and previous assessments. Duration of response: the time from the first documentation of CR or PR or SD to objective disease progression (PD) or death from any cause.
Objective Response Rate (ORR) | up to 5 years after the first patient randomized
  At each visit subjects will be programmatically assigned a RECIST visit response of CR, PR, SD or PD depending on the status of their disease compared to baseline and previous assessments. Objective response rate: the percentage of subjects who have at least one visit response of CR or PR prior to any evidence of progression .
Progression Free Survival（PFS） | up to 5 years after the first patient randomized
  At each visit subjects will be programmatically assigned a RECIST visit response of CR, PR, SD or PD depending on the status of their disease compared to baseline and previous assessments. Progression Free Survival (PFS) : the time from start of study treatment to the first documentation of objective disease progression (PD) or death from any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Liang_an Chen, MD, phD, Principal Investigator — Chinese PLA General Hospital
Locations (4):
- China (4):
  - Chinese PLA General Hospital, Beijing, Beijing Municipality
  - Affiliated hospital of Shandong University of traditional Chinese medicine, Jinan, Shandong
  - Shandong Provincial Hospital, Jinan, Shandong
  - Xijing Hospital affiliated to the Fourth Military Medical University, Xi’an, Shanxi

IPD SHARING:
Plan to Share IPD: No
Because of personal privacy, the research-related individual participant data do not intend for public sharing.

REFERENCES:
- [Derived] Zhu M, Yang Z, Yu H, Zhu Q, Xu Y, Li Y, Li C, Zhao W, Liang Z, Chen L. The efficacy and safety of low-frequency rotating static magnetic field therapy combined with chemotherapy on advanced lung cancer patients: a randomized, double-blinded, controlled clinical trial. Int J Radiat Biol. 2020 Jul;96(7):943-950. doi: 10.1080/09553002.2020.1748737. Epub 2020 Apr 13. PMID 32238091